CLINICAL TRIAL: NCT07125482
Title: Abdominal Massage Group Bed Exercise Group Control Group
Brief Title: Effect of Abdominal Massage and Bed Exercise on Palliative Care Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, SERAP GÜNGÖR ÜNAL, PhD Lecturer, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Abdominal massage
Record Dates: First submitted 2025-05-25; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-06

CONDITIONS: Gastrointestinal Complication; Palliative Care, Patient Care
Keywords: palliative care; comfort; gastrointestinal complication
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Experimental): - Standard nursing care will be applied to the patient.
  Interventions: Other: control group
- abdominal massage group (Experimental): * In this group, patients will receive abdominal massage by the researcher, in addition to routine care, with privacy.
  * Abdominal massage will be applied to the patient by the researcher every morning between 07-08 and 19-20 for 3 days before enteral feeding, and measurements will be recorded 24 hours after the application at 07-08 in the morning. The timing and frequency of massage application were decided according to studies in the literature and expert opinions (Uysal et al., 2012; Wang et al., 2022; Zhang et al., 2023).
  * Before abdominal massage, the patient will be placed in a supine position and will remain in the same position throughout the procedure.
  * For abdominal massage, superficial effleurage, deep effleurage, petrissage, vibration and superficial effleurage maneuvers will be applied to the patient for approximately 15 minutes, respectively.
  * After the application, the patient will be placed in a semi-fawler position
  Interventions: Other: abdominal massage
- bed exercise group (Experimental): The in-bed exercise application will be applied to the patient by the researcher every morning between 07-08 for 3 days before enteral feeding and the measurements will be recorded 24 hours after the application.
  The patient will be placed in a supine position before the in-bed exercise application and will be kept in the same position throughout the procedure.
  For the in-bed exercise application, the following will be applied to the patient, in order; opening and closing the wrist and fingers inwards and outwards, opening and closing the elbow and arm, turning the arm right and left at the level of the head, ankle up and down and right and left, bending and releasing the hip and knee, opening and closing the leg sideways, pushing and pulling the hip and knee 90°, and leg up and down movements will be applied for approximately 15 minutes.
  After the application, the patient will be placed in the semi-fawler position.
  Interventions: Other: bed exercise group

INTERVENTIONS:
Other: bed exercise group — In the first interview, demographic data and other patient information will be collected from the patient record file between 07-08 in the morning before starting bed exercise and nutrition, and the "Patient Information Form" and "Comfort Behavior Checklist, Wong-Baker Face Pain Scale", 'Enteral Nutrition Monitoring Form' will be filled in by the researcher before the intervention and nutrition (1st Interview).
  * In the first interview, bed exercises will be applied by the researcher for approximately 15 minutes before nutrition between 07-08 in the morning (1st Interview).
  * In the second interview, bed exercises will be repeated for approximately 15 minutes after filling out the 'Enteral Nutrition Monitoring Form' before bed exercise and nutrition between 07-08 in the morning (2nd Interview).
  * In the third interview, bed exercises will be repeated for approximately 15 minutes after filling out the 'Enteral Nutrition Monitoring Form' before bed exercise and nutrition between 07-08 in
  Arms: bed exercise group
Other: abdominal massage — * In the first interview, between 07-08 in the morning, demographic data and other information about the patients will be collected from the patient record file before the intervention and feeding by the researcher using the "Patient Information Form" and "Comfort Behavior Checklist, Wong-Baker Facial Pain Scale", 'Enteral Feeding Monitoring Form' (Interview 1).
  * In the first interview, between 07-08 in the morning, abdominal massage will be applied to the patient by the researcher for approximately 15 minutes before feeding (Interview 1).
  * In the second interview, between 07-08 in the morning, abdominal massage will be repeated for approximately 15 minutes by filling out the 'Enteral Feeding Monitoring Form' before feeding and abdominal massage will be repeated (Interview 2).
  * In the third interview, between 07-08 in the morning, the 'Enteral Nutrition Monitoring Form' will be filled out before abdominal massage and feeding, and the abdominal massage will be repeated for approxim
  Arms: abdominal massage group
Other: control group — In the first interview, between 07-08 am, demographic data and other patient information will be collected from the patient record file before feeding, using the "Patient Information Form" and the "Comfort Behavior Checklist, Wong-Baker Facial Pain Scale", 'Enteral Feeding Monitoring Form', before the intervention and feeding (Interview 1).
  * In the second interview, between 07-08 am, the 'Enteral Feeding Monitoring Form' will be filled out before feeding (Interview 2).
  * In the third interview, between 07-08 am, the 'Enteral Feeding Monitoring Form' will be filled out before feeding (Interview 3).
  * In the fourth interview, between 07-08 in the morning, data will be collected with the "Comfort Behavior Checklist", Wong-Baker Facial Pain Scale and 'Enteral Feeding Monitoring Form' before feeding (Interview 4).
  Arms: control group

SUMMARY:
Palliative care is a special type of medical care that focuses on providing support and improving the quality of life for individuals facing life-threatening illnesses. Nursing care for patients receiving enteral nutrition includes interventions that facilitate nutrition, increase patient comfort, and reduce complications. This study will be conducted as a randomized controlled experimental study to evaluate the effects of abdominal massage and in-bed exercise on gastrointestinal complications and patient comfort in palliative care patients.

DETAILED DESCRIPTION:
Abdominal Massage Group Application Steps

* In this group, patients will receive abdominal massage by the researcher in addition to routine care, with privacy provided.
* Abdominal massage will be applied to the patient by the researcher every morning between 07-08 and 19-20 for 3 days before enteral feeding, and measurements will be recorded 24 hours after the application at 07-08 in the morning. The timing and frequency of massage application were decided according to studies in the literature and expert opinions.
* Before abdominal massage, the patient will be placed in a supine position and will remain in the same position throughout the procedure.
* For abdominal massage, superficial effleurage, deep effleurage, petrissage, vibration, and superficial effleurage maneuvers will be applied to the patient for approximately 15 minutes, respectively.
* After the application, the patient will be placed in a semi-fawler position. In-bed Exercise Group Application Steps In-bed exercise application will be applied to the patient by the researcher every morning between 07-08 for 3 days before enteral feeding and measurements will be recorded 24 hours after the application.

Before the in-bed exercise application, the patient will be placed in a supine position and will be kept in the same position throughout the procedure.

For the in-bed exercise application to the patient; opening and closing the wrist and fingers inwards and outwards, opening and closing the elbow and arm, turning the arm right and left at the level of the head, ankle up and down and right and left, bending and releasing the hip and knee, opening and closing the leg sideways, pushing and pulling the hip and knee 90 ͦ, and leg movements in the up and down direction will be applied for approximately 15 minutes.

After the application, the patient will be placed in the semi-fawler position. Control Group Application Steps

* Standard nursing care will be applied to the patient. Abdominal massage group
* In the first interview, between 07-08 in the morning, abdominal massage and demographic data before feeding and other information about the patients will be filled in by the researcher from the patient record file, "Patient Information Form" and "Comfort Behavior Checklist, Wong-Baker Face Pain Scale", 'Enteral Feeding Monitoring Form' before the intervention and feeding (1st Interview).
* In the first interview, between 07-08 in the morning, abdominal massage will be applied to the patient by the researcher for approximately 15 minutes before feeding (1st Interview).
* In the second interview, between 07-08 in the morning, abdominal massage and 'Enteral Feeding Monitoring Form' will be filled in before feeding and abdominal massage will be repeated for approximately 15 minutes (2nd Interview).
* In the third interview, between 07-08 in the morning, abdominal massage and 'Enteral Feeding Monitoring Form' will be filled in before feeding and abdominal massage will be repeated for approximately 15 minutes (3rd Interview).
* In the fourth interview, between 07-08 in the morning, data will be collected with the "Comfort Behavior Checklist", "Wong-Baker Facial Pain Scale" and 'Enteral Nutrition Monitoring Form' before feeding (4th Interview).

In-bed exercise group

* In the first interview, between 07-08 in the morning, demographic data and other information about the patients will be collected from the patient record file before starting the in-bed exercise and feeding, and the "Patient Information Form" and "Comfort Behavior Checklist, Wong-Baker Facial Pain Scale", 'Enteral Nutrition Monitoring Form' will be filled out by the researcher before the intervention and feeding (1st Interview).
* In the first interview, between 07-08 in the morning, in-bed exercises will be applied by the researcher for approximately 15 minutes before feeding (1st Interview).
* In the second interview, between 07-08 in the morning, the 'Enteral Nutrition Monitoring Form' will be filled out before the in-bed exercise and feeding and the in-bed exercises will be repeated for approximately 15 minutes (2nd Interview).
* In the third interview, between 07-08 in the morning, the 'Enteral Nutrition Monitoring Form' will be filled in before bed exercise and feeding, and the in-bed exercises will be repeated for approximately 15 minutes (3rd Interview).
* In the fourth interview, between 07-08 in the morning, the Comfort Behavior Checklist, Wong-Baker Facial Pain Scale and 'Enteral Nutrition Monitoring Form' will be collected before feeding (4th Interview).

Control group

* In the first interview, between 07-08 in the morning, demographic data and other information about the patients will be collected from the patient record file by the researcher before feeding, the "Patient Information Form" and the "Comfort Behavior Checklist, Wong-Baker Facial Pain Scale", 'Enteral Nutrition Monitoring Form' will be filled in before the intervention and feeding (1st Interview).
* In the second interview, between 07-08 in the morning, the 'Enteral Nutrition Monitoring Form' will be filled in before feeding (2nd Interview).
* In the third meeting, between 07-08 am, the 'Enteral Nutrition Monitoring Form' will be filled out before feeding (3rd Meeting). - In the fourth meeting, between 07-08 am, data will be collected with the "Comfort Behavior Checklist", Wong-Baker Facial Pain Scale and 'Enteral Nutrition Monitoring Form' before feeding (4th Meeting).

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age,
* Patients receiving inpatient treatment and care in the palliative care unit,
* Patients who started enteral feeding at least 24 hours ago
* Patients without wounds in the extremity and abdominal region
* Patients without intestinal obstruction
* Patients who have not received abdominal radiotherapy and have not undergone abdominal surgery in the last six weeks
* Patients with a Glasgow Coma Score (GCS) >3
* Patients who have no restrictions on abdominal massage
* Patients whose consent has been obtained from their relatives will be included.

Exclusion Criteria:

* Patients whose enteral feeding was stopped during the study
* Patients who showed signs of infection due to Ventilator-associated Pneumonia or other infections during or before the study will not be included.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
The effect of abdominal massage on gastrointestinal complications | 96 hours
  Abdominal massage was repeated for 3 days, and , diarrhea status and number, constipation status, vomiting status and number, nausea status, abdominal distension, and defecation number measurement were recorded before each abdominal massage.

SECONDARY OUTCOMES:
Effects of in-bed exercise on gastrointestinal complications | 96 hours
  Effects of in-bed exercise was repeated for 3 days, and, diarrhea status and number, constipation status, vomiting status and number, nausea status, abdominal distension, and defecation number measurement were recorded before each in bed exercise.

OTHER OUTCOMES:
The effect of abdominal massage on patient comfort | 96 hours
  The Comfort Behavior Checklist (CBC) consists of 30 behavioral indicators, pain, and comfort scores. The minimum score is 25, and the maximum is 100. Higher scores indicate higher comfort levels. Scoring was done performed before and after the abdominal massage.
The effect of in-bed exercise on patient comfort | 96 hours
  The Comfort Behavior Checklist (CBC) consists of 30 behavioral indicators, pain, and comfort scores. The minimum score is 25, and the maximum score is 100. Higher scores indicate higher levels of comfort. Scoring was done before and after starting in-bed exercises.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaras Sutcu Imam Unıversity, Kahramanmaraş, Kahramanmaraş, Turkey (Türkiye)